CLINICAL TRIAL: NCT03516994
Title: REducing Disparities in the QUALity of Palliative Care for Older African Americans Through Improved Advance Care Planning (EQUAL ACP)
Brief Title: Reducing Disparities in the Quality of Advance Care Planning for Older Adults
Acronym: EQUALACP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00091633; OLC-1609-36381 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2018-04-30; First posted 2018-05-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Cancer; Congestive Heart Failure; Chronic Obstructive Pulmonary Disease; Parkinson Disease; Interstitial Lung Disease; Amyotrophic Lateral Sclerosis; End Stage Liver Disease; End Stage Renal Disease; Diabetes Complications
Keywords: Advance Care Planning; Disparities; Palliative Care; End of Life Care; African Americans
MeSH Terms: conditions — Neoplasm Metastasis; Heart Failure; Pulmonary Disease, Chronic Obstructive; Parkinson Disease; Lung Diseases, Interstitial; Amyotrophic Lateral Sclerosis; End Stage Liver Disease; Kidney Failure, Chronic; Diabetes Complications

STUDY DESIGN:
Intervention Model Description: Mixed-methods, longitudinal, multi-site study, cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Advance Care Planning (Experimental): In the structured advance care planning approach, patients will participate in a 60 to 90 minute facilitated advance care planning conversation with a trained person using Respecting Choices (First Steps) guide and will receive a state advance directive form. The advance care planning facilitator will follow-up as needed after the session to answer additional questions.
  Interventions: Behavioral: Respecting Choices First Steps
- Patient Driven Advance Care Planning (Active Comparator): In the patient-driven advance care planning approach, patients receive a Five Wishes Form (easy to understand advance directive written in plain language), a state advance directive form, and at least two follow-up phone calls with an advance care planning contact who will answer questions.
  Interventions: Behavioral: Five Wishes Form

INTERVENTIONS:
Behavioral: Respecting Choices First Steps — Advance Care Planning Approach
  Arms: Structured Advance Care Planning
Behavioral: Five Wishes Form — Advance Care Planning Approach
  Arms: Patient Driven Advance Care Planning

SUMMARY:
This study compares the effectiveness of two different approaches to advance care planning among older African Americans and older Whites living in the community. The two approaches are a structured approach with an advance care planning conversation led by a trained person using Respecting Choices (First Steps) and a patient-driven approach which includes a Five Wishes advance care planning form written in plain language. The study will determine which approach is more effective at increasing advance care planning within each racial group and reducing differences between the two groups in advance care planning.

DETAILED DESCRIPTION:
Advance care planning (ACP) involves patients making decisions about the kind of medical care they would want to receive if they became unable to speak for themselves. Patients share their wishes in a written document (living will or healthcare proxy) and/or discuss their wishes with family, friends, and doctors. ACP improves the quality of end-of-life care by increasing the likelihood that patients receive care that reflects their preferences and values. Seriously ill African Americans are less likely to take part in advance care planning and experience lower quality care at the end of life, including poorer communication with clinicians and a lower likelihood of receiving the kind of care that they would want.

This study will include 800 seriously or chronically ill community-dwelling older adults (equal number of African Americans and whites) and their caregivers from 10 primary care practices at five medical centers in the Deep South. Eligible patients include those with cancer, advanced heart disease, advanced lung disease, end-stage kidney disease, cirrhosis, diabetes with severe complications, recurrent hospitalizations, or difficulty with basic activities of daily living. For each enrolled patient, one caregiver who is likely to assist the patient with healthcare decisions is also eligible to participate.

The goals of the study are to:

* Compare the effectiveness of two approaches to increasing formal advance care planning (completing written documents like living wills, health care proxies, medical orders for life-sustaining treatments, or other advance directives) and informal advance care planning (having conversations with doctors, family, friends, and others about wishes for future healthcare) for African Americans and for Whites.
* Determine which intervention is most effective in reducing differences between African Americans and Whites in rates of advance care planning.
* Determine whether the effectiveness of the advance care planning approach differs based on whether the person assisting with advance care planning is of the same or different race as the patient.

Administered by community health workers, the two advance care planning approaches which will be compared are:

* Patient-driven approach which includes a Five Wishes Form (advance directive written in easy to understand language)
* Structured approach with an advance care planning conversation led by a trained person using Respecting Choices (First Step) conversation guide.

ELIGIBILITY:
Inclusion Criteria for Patients:

* African-American or White
* age 65 or greater
* English-speaking
* residing in non-institutional setting
* cognitively able to participate in advance care planning
* Serious or chronic illness including: metastatic cancer; end stage renal disease; advanced liver disease, heart disease or lung disease; amyotrophic lateral sclerosis, severe Parkinson's disease; 2 or more unplanned hospitalizations in the last year; requiring assistance with any basic activity of daily living
* Serious illness based on the following: Clinician answers "no" to the surprise question: "Would you be surprised if this person died in the next 12 months?"

Exclusion Criteria for Patients:

* residence in nursing home or assisted living facility
* diagnosis of dementia or unable to consent
* documented advance care plan (living will, health care proxy, MOST form, provider note)
* current or prior use of hospice
* current or prior use of non-hospice palliative care except inpatient palliative care consultation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 790 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Proportion of African Americans who complete advance care planning | 12 months
  completion of an advance care planning document (living will, healthcare proxy, medical orders, Five Wishes, other); discussion with clinician documented in chart, patient report of advance care planning discussion (designated decision-maker, discussed values, goals, preferences) with family, friends, or others
Proportion of Whites who complete advance care planning | 12 months
  completion of an advance care planning document (living will, healthcare proxy, medical orders, Five Wishes, other); discussion with clinician documented in chart, patient report of advance care planning discussion (designated decision-maker, discussed values, goals, preferences) with family, friends, or others

SECONDARY OUTCOMES:
Difference in Proportion of Whites versus African Americans who complete advance care planning | 12 months
  Difference of proportion in whites versus African Americans who complete formal or informal advance care planning
Patient Readiness to Engage in Advance Care Planning | 3 months
  Measure assessing patient's readiness to name decision-maker, discuss care preferences, complete legal advance directive
Patient Quality of Life | 3 months, 6 months, one year
  Measure (Promis 29) assessing quality of life, including domains of physical functional, emotional, and social well-being

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Johnson, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Emory University, Atlanta, Georgia
  - University of South Carolina, Columbia, South Carolina
  - University of Texas Southwestern, Dallas, Texas